CLINICAL TRIAL: NCT05068765
Title: The Effect of Communication Skills Focused Psychoeducation on Subjective Well-Being of the Caregivers of Individual With the Diagnosis of Schizophrenia
Brief Title: The Effect of the Psychoeducation Program on the Subjective Well-being of Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ŞİRİN HARKİN (Other)
Responsible Party: Sponsor-Investigator, ŞİRİN HARKİN, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 157435
Record Dates: First submitted 2021-08-02; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Caregiver; Psychoeducation; Communication Skills; Well-being
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Once enrolled and consent is documented, eligible subject's will participate in the study for approximately six months.
- communication skills psychoeducation (Experimental): Communication skills focused psychoeducation group will be given a communication skills-focused psychoeducation program for eight weeks, one session per week, for a total of eight sessions. The number of sessions was planned with reference to the study in which the effect of the psychoeducation program on general health and communication skills in caregivers of individuals with schizophrenia was investigated.Session groups will be formed from a single session of 60-90 minutes for each topic.
  Interventions: Other: Communication skills psychoeducation
- general psychoeducation (Experimental): General psychoeducation group will be given a general psychoeducation program for four weeks, one session per week, in total. Session groups will be formed from a single session of 60-90 minutes for each topic.
  Interventions: Other: General psychoeducation

INTERVENTIONS:
Other: Communication skills psychoeducation — Intervention explanations are explained in the groups section.
  Arms: communication skills psychoeducation
Other: General psychoeducation — İntervention descriptions are explained in the intervention groups section.
  Arms: general psychoeducation

SUMMARY:
This study aims to evaluate the effectiveness of a communication skills-focused psychoeducation program on the subjective well-being of primary caregivers of individuals with schizophrenia.

Today, with the adoption of contemporary treatment models, the relatives of individuals with schizophrenia have become caregivers. Some caregivers who are not competent enough to communicate satisfactorily with a person diagnosed with schizophrenia may have problems in patient-patient-relative interaction. Problems that occur frequently in expressing oneself, giving appropriate reactions in interaction with the patient and creating a sense of trust are seen as a major source of concern by caregivers. In the solution of this problem, improving the communication skills of the caregiver and increasing the self-confidence and motivation to communicate with the individual diagnosed with schizophrenia is an area that should be addressed by mental health professionals.

By using a communication skills focused psychoeducation program, it is aimed to increase the level of subjective well-being of caregivers of individuals with schizophrenia by establishing healthy and positive relationships, coping with the negative emotions and difficulties they face, realizing their strengths, and leading a happy and meaningful life. Within the scope of this aim, it was aimed to evaluate the effect of a communication skills focused psychoeducation program on the subjective well-being of caregivers of individuals with schizophrenia.

DETAILED DESCRIPTION:
This study was planned as an experimental study with a randomized control group in order to evaluate the effect of psychoeducation focused on communication skills on the subjective well-being of caregivers of individuals with schizophrenia.

The population of the research will be family members who apply to ZBEÜ Application and Research Center Psychiatry Outpatient Clinic and care for individuals diagnosed with schizophrenia according to DSM-5 TR criteria. Statistical power analysis was applied for the number of samples. While calculating the power values, the results were determined within the scope of 95% confidence level. According to the power values obtained from the reference study in parallel with the research to be carried out, if this study is studied with a total of 60 observations, a test power of approximately 88.5% is reached. As a result, according to the power analysis, it was determined that the research could be done with 60 observations. The caregiver family members included in the study will be stratified according to the scores they get from the care burden and communication skills scale and some individual characteristics, and an equal number of individuals from each stratum will be selected, and they will be included in two intervention groups and a control group by randomization.

The Criteria for Inclusion of Caregivers in the Research are as follows:

* The patient receiving care should have been diagnosed with schizophrenia at least one year ago according to the DSM-V TR diagnostic criteria,
* Living together with the caregiver for at least six months,
* Being directly (fully) responsible for the care of the patient being cared for,
* Being 18 years or older,
* Residing in the city center of Zonguldak,
* To be at least primary school graduate,
* No hearing and comprehension problems. The first measurements (Information Form, Zarit Care Burden Scale, Subjective Well-Being Scale and Communication Skills Scale) will be collected by making face-to-face preliminary interviews with the caregivers who meet the research criteria and agree to participate in the research.

After the pre-test, intervention and control groups will be formed in line with homogeneity in terms of scale scores and some individual characteristics.

While the control group continues their routine follow-ups, psychoeducation focused on communication skills will be applied to the first intervention group and general psychoeducation program to the second intervention group.

After the psychoeducation program is completed, final measurements will be collected for intervention and control groups. Follow-up measurements will be made in the intervention and control groups in the 1st and 3rd months.

The first intervention group will be given a communication skills-focused psychoeducation program for eight weeks, one session per week, for a total of eight sessions. The number of sessions was planned with reference to the study in which the effect of the psychoeducation program on general health and communication skills in caregivers of individuals with schizophrenia was investigated. The second intervention group will be given a general psychoeducation program for four weeks, one session per week, in total. Session groups will be formed from a single session of 60-90 minutes for each topic.

Scales Subjective well-being scale: The scale is a five-point Likert type consisting of 46 items. The aim of the scale is to determine the subjective well-being levels of individuals by determining the frequency and intensity of positive and negative emotions with their cognitive evaluations of their lives. Subjective well-being scale consists of personal judgments and positive and negative emotional expressions about living spaces. The lowest score that can be obtained from the scale is 46, and the highest score is 230. A high score indicates a high level of subjective well-being.

ELIGIBILITY:
Inclusion Criteria:

* The patient receiving care has a diagnosis of schizophrenia,
* Living with the patient receiving care for 6 months,
* Being directly (full) responsible for the care of the patient being cared for,
* Be over 18 years old,
* Living in the city center of Zonguldak,
* To be at least primary school graduate,
* Having no hearing and comprehension problems,

Exclusion Criteria:

• Having a history of substance abuse (excluding nicotine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of the "subjective well-being scale" score averages of the participants in the communication skills psychoeducation group before and after the training | 12 months
  After the 8-week training program was applied to the communication skills psychoeducation group, it is expected that the subjective well-being scale scores of the participants will increase. Subjective well-being scale data will be collected before and after the training. The scale will be repeated one month and three months after training. Subjective well-being scale consists of personal judgments and positive and negative emotional expressions about living spaces. The lowest score that can be obtained from the scale is 46, and the highest score is 230. A high score indicates a high level of subjective well-being. Quantitative data will be used to measure the change in participants' views and feelings before and after the training. The data will be analyzed using the Statistical Package for Social Sciences package program.
The change of the "subjective well-being scale" mean scores of the participants in the communication skills psychoeducation group after the training compared to the mean scores of the control group participants | 12 months
  After the training, the difference in the "subjective well-being scale" score averages of the communication skills psychoeducation and control group participants will be examined.After the 8-week training program was applied to the communication skills psychoeducation group, it is expected that the subjective well-being scale mean scores of the participants will increase compared to the control group.Control group participants will not receive any intervention. Subjective well-being scale data will be collected before and after the training. The scale will be repeated one month and three months after the training. Subjective well-being scale consists of personal judgments and positive and negative emotional expressions about living spaces. The lowest score that can be obtained from the scale is 46, and the highest score is 230. A high score indicates a high level of subjective well-being.
The change of the "subjective well-being scale" score averages of the communication skills focused psychoeducation group participants after the training compared to the general psychoeducation group participants' mean scores | 12 months
  After the training, the difference between the subjective well-being scale scores of the participants in the communication skills psychoeducation group and the scores of the participants in the general psychoeducation group will be examined. It is expected that the mean scores of the communication skills psychoeducation group will be higher than the general psychoeducation group. An 8-week training program will be applied to the communication skills focused psychoeducation group, and a general psychoeducation program will be applied to the general psychoeducation group. Subjective well-being scale data will be collected before and after the training. The scale will be repeated one month and three months after the training. The lowest score that can be obtained from the scale is 46, and the highest score is 230.A high score indicates a high level of subjective well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Bilgin, Prof., Study Director — Istanbul University-Cerrahpasa Florence Nightingale Nursing Faculty Mental Health and Psychiatric Nursing Department
Locations (1):
- Zonguldak Bulent Ecevit University Health Practice and Research Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months

REFERENCES:
- [Background] Gharavi Y, Stringer B, Hoogendoorn A, Boogaarts J, Van Raaij B, Van Meijel B. Evaluation of an interaction-skills training for reducing the burden of family caregivers of patients with severe mental illness: a pre-posttest design. BMC Psychiatry. 2018 Mar 27;18(1):84. doi: 10.1186/s12888-018-1669-z. PMID 29587690
- See also: Rezaei, et al. (2018). Applying psychoeducational program on general health and communication skills in caregivers of patients with schizophrenia: a randomized controlled trial. The European Journal of Psychiatry, 32(4), 174-181 — https://doi.org/10.1016/j.ejpsy.2018.04.001